CLINICAL TRIAL: NCT03620721
Title: Effectiveness and Implementation of a Mindfulness Intervention for Depressive Symptoms Among Low-income, Racial/Ethnic Minority Adults in a Federally Qualified Health Center
Brief Title: Effectiveness and Implementation of a Mindfulness Intervention for Depressive Symptoms Among Adults in a FQHC
Acronym: M-Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Inger Burnett-Zeigler, Assosciate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00207126
Record Dates: First submitted 2018-07-23; First posted 2018-08-08 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Depressive Symptoms; Stress, Psychological; Stress, Physiological
MeSH Terms: conditions — Depression; Stress, Psychological | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-Body (Experimental): mindfulness group intervention
  Interventions: Behavioral: mindfulness
- Usual Care (No Intervention): treatment as usual

INTERVENTIONS:
Behavioral: mindfulness — 8-week mindfulness based group intervention
  Arms: M-Body

SUMMARY:
The objective of this project is to examine the clinical effectiveness of a mindfulness intervention on reducing depressive symptoms among socio-economically disadvantaged, racial/ethnic minority adults and explore factors related to implementation in a Federally Qualified Health Center (FQHC). This research will be used to develop a generalizable model for delivery of streamlined mental health interventions in community based settings that will be broadly disseminated and scalable to other populations. Black and Hispanic adults are more likely than those who are White to receive depression treatment in primary care, where antidepressants are the most commonly offered treatment. However, Black and Hispanic adults are less likely than Whites to find antidepressants acceptable. A mindfulness depression intervention provided within primary care may be more accessible and acceptable for low-income, racial/ethnic minority individuals, a severely underserved population. The investigators will conduct a randomized controlled trial to test the clinical effectiveness of a mindfulness intervention (M-Body) on reducing depressive symptoms, compared to usual care, among low-income racial/ethnic minority adults in a FQHC. The M-Body intervention is based on Mindfulness Based Stress Reduction and has been tailored for the FQHC setting and patient population. Adults (N=254) with depressive symptoms will be recruited from a FQHC in the Chicago, IL area that serves majority racial/ethnic minority individuals (90%) living at or below the poverty line (74%). Half of the patients will be randomized to the M-Body intervention arm where they will receive 8-weeks of mindfulness training led by FQHC staff and the other half will be randomized to usual care. Information on factors relevant to implementation of the intervention in the FQHC will be obtained by convening a series of workgroups and individual interviews with FQHC staff, executive leadership and community stakeholders. Specific Aims: 1) Determine the effectiveness of M-Body on reducing depressive symptoms compared to enhanced usual care for racial/ethnic minority adults in a FQHC; 2) Explore potential mediators (stress related biomarkers, mindfulness) and moderators (age, personal, social, environmental stressors) of the intervention's effect; 3) Conduct a broad assessment of organizational and individual agency factors related to preparation and implementation of the M-Body intervention in a FQHC using a mixed methods approach.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* mild to severe depressive symptoms (Patient Health Questionnaire-9, PHQ-9, total score ≥ 5)
* English speaking

Exclusion Criteria:

* PHQ-9 total score <5
* past 30-day suicidal ideation
* current, regular practice of meditation (≥ 4 per week)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms | 6 months
  Inventory of Depressive Symptoms (IDS-C), 30 items rated on a 0-3 point scale, total scores range from 0-84

SECONDARY OUTCOMES:
Anxiety | 6 months
  Generalized Anxiety Disorder (GAD-7), 7 items, rated on a 0-3 point scale
Anger | 6 months
  Anger Self-Report Questionnaire (ASRQ), 30 items rated on a 1-6 point scale

OTHER OUTCOMES:
Self-reported Stress | 6 months
  Perceived Stress Scale (PSS), 10 items rated on a 0-4 point scale
Mindfulness | 6 months
  Five Facet Mindfulness Questionnaire (FFMQ), 14 items rated on a 1-5 point scale
Cognitive Reactivity | 6 months
  Cognitive Emotion Regulation Questionnaire (CERQ), 36 items rated on a 1-5 point scale
Self-Compassion | 6-months
  Self Compassion Scale (SCS), 26 items rated on a 1-5 point scale
Affective Dysregulation | 6 months
  Difficulties in Emotion Regulation Scale (DERS), 36 items rated on a 1-5 point scale
Negative Thinking | 6 months
  Reflection and Rumination Questionnaire (RRQ), 24 items rated on a 1-5 point scale
Social Functioning | Baseline
  Social Problems Questionnaire (SPQ), 33 items rated on a 0-3 point scale
Traumatic Life Events | 6 months
  PTSD Checklist for DSM-5 (PCL-5) with Life Events Checklist-5 (LEC-5), 20 items rated on a 0-4 point scale with an additional 17 items checklist
Spirituality | Baseline
  Spirituality Scale (SS), 8 items rated on a 1-6 point scale
Blood Pressure | Baseline, 8, 16, and 24 weeks
  Ranges of blood pressure measurements (mmHg)
Inflammatory Biomarkers | Baseline, 8, 16, and 24 weeks
  Dried Blood Spot (DBS) samples will be assessed for inflammatory biomarkers (CRP, IL6, and IL8)
Race-Based Stress | Baseline and 8 weeks
  Racial and Ethnic Microaggressions Scale (REMS), 28 items rated on a 0-5 point scale

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Asher Center for the Study and Treatment of Depressive Disorders, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haidar A, Schauer J, Gurra M, Burnett-Zeigler I. The Impact of the COVID-19 Pandemic on Depression, Anxiety, and Stress among Black Women with Depressive Symptoms at a Federally Qualified Health Center. J Racial Ethn Health Disparities. 2025 Jun;12(3):1657-1664. doi: 10.1007/s40615-024-01998-y. Epub 2024 Apr 18. PMID 38635151
- [Derived] Burnett-Zeigler I, Zhou E, Martinez JH, Zumpf K, Lartey L, Moskowitz JT, Wisner KL, McDade T, Brown CH, Gollan J, Ciolino JD, Schauer JM, Petito LC. Comparative effectiveness of a mindfulness-based intervention (M-Body) on depressive symptoms: study protocol of a randomized controlled trial in a Federally Qualified Health Center (FQHC). Trials. 2023 Feb 17;24(1):115. doi: 10.1186/s13063-022-07012-2. PMID 36803835